CLINICAL TRIAL: NCT05519319
Title: Clinical Effect and Safety of Photodynamic Therapy Versus Radiofrequency Ablation Versus Photodynamic Therapy Plus Radiofrequency Ablation for Unresectable Extrahepatic Cholangiocarcinoma
Brief Title: Safety and Efficacy of PDT vs RFA vs PDT+RFA for the Treatment of Extrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, Professor, First People's Hospital of Hangzhou
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-01
Record Dates: First submitted 2022-08-24; First posted 2022-08-29 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Extrahepatic Cholangiocarcinoma; Bile Duct Cancer
Keywords: Extrahepatic cholangiocarcinoma; Photodynamic therapy; Radiofrequency ablation
MeSH Terms: conditions — Cholangiocarcinoma; Bile Duct Neoplasms | interventions — 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Intervention Model Description: Three parallel groups
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessor are unaware about the results
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Photodynamic therapy(PDT) (Active Comparator): The PDT optical fiber was inserted through the dilation catheterand advanced toward the bile duct stenosis point under visual-radiography. The dilation catheter was then withdrawn to leave the PDT optical fiber directly across the stricture. Photoactivation was performed at 640 nm using a diode laser at a light dose of 180 J/cm2at power density of300 mW/cm2 and irradiation time of 600 s.
  Interventions: Procedure: PDT
- Radiofrequency ablation(RFA) (Active Comparator): An RFA electrode (Habib EndoHPB, EMcision, HitchinHerts, UK) was advanced along the guide wire into the bile duct and to the biliary stricture under X-ray fluoroscopic guidance. A 400 kHz RF generator (RITA 1500X, Angio Dynamics, USA) was connected for RFA at 7-10 W for 90 seconds.
  Interventions: Procedure: RFA
- RFA+PDT (Active Comparator): The PDT optical fiber was inserted through the dilation catheterand advanced toward the bile duct stenosis point under visual-radiography. The dilation catheter was then withdrawn to leave the PDT optical fiber directly across the stricture. Photoactivation was performed at 640 nm using a diode laser at a light dose of 180 J/cm2at power density of300 mW/cm2 and irradiation time of 600 s. After that An RFA electrode (Habib EndoHPB, EMcision, HitchinHerts, UK) was advanced along the guide wire into the bile duct and to the biliary stricture under X-ray fluoroscopic guidance. A 400 kHz RF generator (RITA 1500X, Angio Dynamics, USA) was connected for RFA at 7-10 W for 90 seconds.
  Interventions: Procedure: RFA combined with PDT

INTERVENTIONS:
Procedure: RFA — RFA will be performed
  Other Names: ERCP guided
  Arms: Radiofrequency ablation(RFA)
Procedure: PDT — PDT will be performed
  Other Names: ERCP guided
  Arms: Photodynamic therapy(PDT)
Procedure: RFA combined with PDT — RFA and PDT will be performed
  Other Names: ERCP guided
  Arms: RFA+PDT

SUMMARY:
A median survival period of 3 to 6 months is the prognosis for patients with advanced, unresectable EHCC. For patients with locally advanced, unresectable EHCC, effective management of tumor growth is the only option to increase stent patency and survival time. In patients with cholangiocarcinoma, photodynamic therapy (PDT) is therapy that has been shown to improve stent patency and overall survival (OS). Endoscopic radiofrequency ablation (RFA) has been demonstrated in numerous studies to prolong the life spans of individuals with malignant biliary obstruction . In the literature, comparing the clinical efficacy and adverse outcomes of these two endoscopic procedures is rare.

DETAILED DESCRIPTION:
The lower common bile duct and the hepatic hilar area are the origin of extrahepatic cholangiocarcinoma (EHCC). Patients with advanced, unresectable EHCC have a relatively poor prognosis, with a median survival time of 3 to 6 months. The only way to prolong stent patency and survival for patients with unresectable locally advanced EHCC is by active control of tumor development. The only treatment that has consistently demonstrated an improvement in stent patency and overall survival (OS) in cholangiocarcinoma patients is photodynamic therapy (PDT). The popularity of endoscopic retrograde cholangio-pancreatography (ERCP)-guided radiofrequency ablation (RFA) has grown recently in an effort to increase stent patency and survival time for patients with malignant biliary obstruction.RFA for biliary cholangiocarcinoma has demonstrated safety and effectiveness. Endoscopic RFA has been shown in various studies to prolong stent patency and the survival of patients with malignant biliary obstruction. The clinical effectiveness and adverse events of these two endoscopic treatments have not been compared in many papers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed cholangiocarcinoma;
* unresectable cholangiocarcinoma due to local infiltration of major vessels according to computed tomography (CT), magnetic resonance cholangiopancreatography (MRCP), or endoscopic ultrasound（EUS）;
* No previous treatment;
* Adequate bone marrow and organ function (white blood cells>4.0×109/L, hemoglobin>90 g/L, and platelets>75×109/L, serum creatinine<2.0 mg/dl);
* A Karnofsky performance status (KPS) score ≥ 50;
* Signed written informed consent.

Exclusion Criteria:

* Imaging examination (CT, MRCP, EUS) showed distant metastasis of liver, lung and other organs;
* Coexistent with other malignant tumors;
* Pregnant or nursing women;
* Previous gastrointestinal diversion;
* Participation in another study during the month before enrollment in this study;
* Alcohol and/or substance abuse or potentially poor compliance per a doctor's judgment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Three years
  OS was defined as the time from initial RFA or PDT to death or the end of the study.

SECONDARY OUTCOMES:
Adverse events | Three years
  Number of patients with adverse events
Progression-free survival(PFS) | Three years
  PFS was measured from therapy until the date of disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhang, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Yet not decided

REFERENCES:
- [Background] Gao DJ, Yang JF, Ma SR, Wu J, Wang TT, Jin HB, Xia MX, Zhang YC, Shen HZ, Ye X, Zhang XF, Hu B. Endoscopic radiofrequency ablation plus plastic stent placement versus stent placement alone for unresectable extrahepatic biliary cancer: a multicenter randomized controlled trial. Gastrointest Endosc. 2021 Jul;94(1):91-100.e2. doi: 10.1016/j.gie.2020.12.016. Epub 2020 Dec 24. PMID 33359435
- [Result] Chen P, Yang T, Shi P, Shen J, Feng Q, Su J. Benefits and safety of photodynamic therapy in patients with hilar cholangiocarcinoma: A meta-analysis. Photodiagnosis Photodyn Ther. 2022 Mar;37:102712. doi: 10.1016/j.pdpdt.2022.102712. Epub 2022 Jan 5. PMID 34995788
- [Result] Li Z, Jiang X, Xiao H, Chen S, Zhu W, Lu H, Cao L, Xue P, Li H, Zhang D. Long-term results of ERCP- or PTCS-directed photodynamic therapy for unresectable hilar cholangiocarcinoma. Surg Endosc. 2021 Oct;35(10):5655-5664. doi: 10.1007/s00464-020-08095-1. Epub 2020 Oct 26. PMID 33104917
- [Result] Yang J, Wang J, Zhou H, Zhou Y, Wang Y, Jin H, Lou Q, Zhang X. Efficacy and safety of endoscopic radiofrequency ablation for unresectable extrahepatic cholangiocarcinoma: a randomized trial. Endoscopy. 2018 Aug;50(8):751-760. doi: 10.1055/s-0043-124870. Epub 2018 Jan 17. PMID 29342492